CLINICAL TRIAL: NCT01834885
Title: A 12-week Treatment, Multi-center, Randomized, Double-blind, Double-dummy, Parallel-group Study to Assess the Efficacy, Safety and Tolerability of QVA149 Compared to Fluticasone/Salmeterol in COPD Patients With Moderate to Severe Airflow Limitation
Brief Title: A 12 Week Study of QVA149 Compared to Fluticasone/Salmeterol (Advair) for Treatment of COPD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQVA149A2327
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol-glycopyrronium combination; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- QVA149 (Experimental): QVA149 study medication kit will contain blister strips and a unique inhaler. Patients will be instructed to inhale their medication twice a day for 12 weeks.
  Interventions: Drug: QVA149
- fluticasone/salmeterol (Active Comparator): Fluticasone/salmeterol study medication kit will contain an inhaler in the manufacturer's device. Patients will be instructed to inhale their medication twice a day for 12 weeks.
  Interventions: Drug: fluticasone/salmeterol

INTERVENTIONS:
Drug: QVA149 — QVA149 via inhaler twice a day
  Arms: QVA149
Drug: fluticasone/salmeterol — fluticasone/slameterol via inhaler twice a day
  Arms: fluticasone/salmeterol

SUMMARY:
Study is to show that QVA149 is superior to the standard of care, fluticasone/salmeterol, in patients with moderate to severe airflow limitation

ELIGIBILITY:
Inclusion Criteria:

* Age >= 40 years, patients with airflow limitation indicated by post-bronchdilation FEV1 >=30% and <80% of predicted normal, current or ex-smokers with a 10 pack year smoking history, patients with a mMRC grade 2 or greater

Exclusion Criteria:

* prolonged QTCF >450 ms, paroxysmal atrial fibrillation, Type I or uncontrolled Type II diabetes, history of asthma, COPD diagnosis before age 40, receiving treatments not allowed in the study, other concomitant pulmonary diseases.

Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) 0-12 hours for FEV1 following 12 weeks of treatment | 12 weeks
  Area under the curve (AUC) 0-12 hours for Forced Expiratory Volume in 1 second (FEV1) following 12 weeks of treatment. AUC will be calculated using the trapezoidal rule and standardized with respect to length of time from the first 5 minute to the last measurement at 12 hours.

SECONDARY OUTCOMES:
Trough Forced Expiratory Volume in 1 second (FEV1) following 12 weeks of treatment | Day 1 and Week 12
  Spiromtery testing conducted according to internationally accepted standards. FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The trough FEV1 will be will be defined as the mean from repeat measurements at Day 1 and week 12.
Transition Dyspnea Index (TDI) Focal Score | Week 12
  Transition Dyspnea Index (TDI) captures changes from baseline. The TDI score is based on three domains with each domain scored from -3 (major deterioration) to +3 (major improvement), to give an overall score of -9 to +9, a negative score indicating a deterioration from baseline. A TDI focal score of 1 is considered to be a clinically significant improvement from baseline; negative scores indicate deterioration. A TDI focal score of 1 unit is considered to be a minimal clinically important difference (MCID) from baseline.
Quality of Lfe Assessment with St George's Respiratory Questionaire (SGRQ) | Week 12
  SGRQ is a health related quality of life questionnaire consisting of 51 items in three components: symptoms, activity, and impacts. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life. Change from baseline in total score will be assessed.
Change from baseline in daily number of puffs of rescue medication | Week 12
  Number of puffs of rescue medication in previous 12 hours is recorded in Patient Diary twice daily. The total number of puffs of rescue medication per day (daily use) over the active treatment period will be used to derive the mean daily number of puffs of rescue medication taken by the patient.
Daily symptoms reported by patient | Week 12
  Patient's daily symptoms will be recorded twice daily using a patient diary. Mean daily total symptom score, mean morning and evening symptom score for each patient will be calculated over the 12 week study period.
COPD assessment (CAT) test | Week 12
  COPD assessment test (CAT) contains 8 questions regarding patient symptoms. Patient will complete questions using a 6 point scale and total score out of a possible score of 40 will be summed and reported.
Safety and tolerability | Over 12 weeks
  All adverse events and serious adverse events (SAEs) will be reported.
Peak Forced Expiratory Volume in 1 second (FEV1) within 4 hours post-dose | Day 1 and Week 12
  Spirometry testing conducted accorded to internationally accepted standards. Peak FEV1 defined as the maximum FEV1 during the first 4 hours post dosing. The Peak FEV1 will be defined as the mean from repeat measurements at Day 1 and week 12.
Area under the curve (AUC) 0-4 hours for FEV1 | Day 1 and Week 12
  Area under the curve (AUC) 0-4 hours for Forced Expiratory Volume in 1 second (FEV1) at Day 1 and week 12. AUC will be calculated using the trapezoidal rule and standardized with respect to length of time from the first 5 minute to the last measurement at 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Austria (6):
  - Novartis Investigative Site, Feldkirch, Austria
  - Novartis Investigative Site, Grieskirchen, Austria
  - Novartis Investigative Site, Hallein, Austria
  - Novartis Investigative Site, Linz, Austria
  - Novartis Investigative Site, Thalheim bei Wels, Austria
  - Novartis Investigative Site, Wels, Austria
- Germany (15):
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Dresden, Germany
  - Novartis Investigative Site, Leipzig, Germany
  - Novartis Investigative Site, Potsdam, Germany
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Rheine